CLINICAL TRIAL: NCT05673694
Title: A Phase Ia/Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of EG017 in Androgen Receptor-positive, Estrogen Receptor-positive, and Human Epidermal Growth Factor Receptor-2-negative Patients With Advanced Breast Cancer.
Brief Title: To Evaluate a Phase Ia/Ib Clinical Study of EG017 in Patients With Advanced Breast Cancer.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EG017
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EG017 (Experimental): 70 subjects: Part Ia 10 subjects: A total of 3 dose groups of 6 mg/day, 18 mg/day, 24 mg/day are planned. Once a day, each treatment cycle was administered for 28 days.
  Part Ib 60 subjects: A total of 2 dose groups of 18 mg/day, 24 or 12mg/day are planned. Once a day, each treatment cycle was administered for 28 days.
  Interventions: Drug: EG017

INTERVENTIONS:
Drug: EG017 — According to the dosage group of the program, once a day.

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics and efficacy of EG017 in androgen receptor-positive, estrogen receptor-positive, and human epidermal growth factor receptor-2-negative patients with advanced breast cancer.

DETAILED DESCRIPTION:
The major aims of the study are to define the safety profile of this new drug, and to determine a recommended.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 18-75 years old;
2. Expected survival ≥ 12 weeks;
3. Subjects with ECOG score of physical state 0~1;
4. Histologically confirmed recurrent or metastatic advanced breast cancer;

Exclusion Criteria:

1. Those who have had a severe allergic reaction to any drug or its components in this study in the past;
2. Present with primary central nervous system (CNS) malignancies; Subjects with CNS metastasis who have failed local treatment (except asymptomatic BMS, or symptomatic BMS with complete remission of symptoms ≥ 2 weeks after treatment for BMS);
3. Has any disease or syndrome that requires or is likely to require systemic steroid therapy during the study period;
4. Gastrointestinal disorders or gastrointestinal diseases will significantly affect the absorption of test drugs (such as ulcerative disease, uncontrolled vomiting, diarrhea, malabsorption syndrome, biliary drainage status, etc.), or subjects cannot take drugs orally:

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal women or women in a postmenopausal state
Enrollment: 70 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-11-07 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of EG017 as Measured by the Number of Participants Experiencing Dose-limiting Toxicities (DLTs), Adverse Events (AEs), and Serious Adverse Events (SAEs). | 28 Days
  The CTCAE criteria will be used to assess adverse events on this trial.
The effectiveness of EG017 in humans was evaluated by clinical benefit rate | 24 Weeks
  The number and proportion of subjects in clinical remission at 24 weeks after administration were calculated

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Cancer Hospital of CAMS, Beijing, Benjing
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan